CLINICAL TRIAL: NCT00623857
Title: Effects of Supplementation With Zinc and Other Micronutrients on the Health and Development of African Children
Brief Title: Micronutrients and Child Health Study
Acronym: MACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WAO 93-442
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Malaria
Keywords: Micronutrients; Zinc; Vitamins; Trace elements; Minerals; Vitamin A; Vitamin B1; Vitamin B2; Niacin; Vitamin B6; Folic acid; Vitamin B12; Vitamin C; Vitamin D; Vitamin E; Vitamin K; Iron; Iodine; Copper; Selenium; Magnesium; Calcium; Malaria; Immunity; Anthropometry
MeSH Terms: conditions — Malaria | interventions — Zinc; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Zinc
  Interventions: Dietary Supplement: Zinc
- 2 (Active Comparator): Vitamins and minerals other than zinc
  Interventions: Dietary Supplement: Vitamins and minerals other than zinc
- 3 (Active Comparator): Vitamins plus zinc and other minerals
  Interventions: Dietary Supplement: Vitamins plus zinc and other minerals
- 4 (Placebo Comparator): Placebo for all vitamins and minerals
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc — Daily oral supplementation with zinc, 10 mg, for an average of 60 weeks
  Arms: 1
Dietary Supplement: Vitamins and minerals other than zinc — Daily supplementation with vitamin A, vitamin B1, vitamin B2, niacin, vitamin B6, folic acid, vitamin B12, vitamin C, vitamin D, vitamin E, vitamin K, iron, iodine, copper, selenium, magnesium and calcium; for an average of 60 weeks
  Arms: 2
Dietary Supplement: Vitamins plus zinc and other minerals — Daily oral supplementation with zinc, vitamin A, vitamin B1, vitamin B2, niacin, vitamin B6, folic acid, vitamin B12, vitamin C, vitamin D, vitamin E, vitamin K, iron, iodine, copper, selenium, magnesium and calcium; for an average of 60 weeks
  Arms: 3
Dietary Supplement: Placebo — Daily oral supplementation with placebo for vitamins and all minerals; for an average of 60 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to determine to what extent supplementation with zinc and other micronutrients are efficacious in preventing malaria in young Tanzanian children.

DETAILED DESCRIPTION:
Zinc is essential for the functioning of the immune system. Supplementation trials in Asia, Latin America, the Pacific and developed countries have shown that increasing zinc intake has great potential to control common infections in children, but the response to supplementation may be different in Africa, where the primary environmental challenge to children's health is malaria. Simultaneous supplementation with other potentially limiting nutrients may be required to overcome a lack of response when zinc is given alone. The project aims at measuring effects of daily oral supplementation with zinc and other micronutrients, given either alone or in combination, on malaria incidence and nutritional status, and on indicators of immunity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-60 months
* Permanently residing in the study area
* Being moderately or mildly stunted (height-for-age z-score <-1.5 SD)
* Informed consent from parents or guardians obtained

Exclusion Criteria:

* Severe wasting (weight-for-height z-score <-3 SD)
* Hemoglobin concentration <70 g/L
* Axillary temperature ≥37.50 °C with malaria antigenemia
* Signs and symptoms at randomisation suggesting malaria, hepatitis, HIV/AIDS, tuberculosis, sickle cell disease or other severe condition
* Unable to produce a venous blood sample (>1 mL)

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 612 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Febrile malaria episodes | 60 weeks

SECONDARY OUTCOMES:
Haematologic and urinary indicators of micronutrient status | 30 weeks after start of intervention
Anthropometric indices | 57 weeks after start of intervention
T cell immune responses to in vitro stimulation with a crude Plasmodium falciparum lysate | 30 weeks after start of intervention
Plasma immunoglobulin concentrations | 2 weeks after malaria episodes

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verhoef, PhD, Principal Investigator — Wageningen University, Cell Biology and Immunology Group; Raimos M Olomi, MD MMed MPH, Study Chair — Kilimanjaro Christian Medical Centre; Huub FJ Savelkoul, PhD, Study Director — Wageningen University, Cell Biology and Immunology Group; John F. Shao, MD, Study Director — Kilimanjaro Christian Medical Centre
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

REFERENCES:
- [Result] Imwong M, Woodrow CJ, Hendriksen IC, Veenemans J, Verhoef H, Faiz MA, Mohanty S, Mishra S, Mtove G, Gesase S, Seni A, Chhaganlal KD, Day NP, Dondorp AM, White NJ. Plasma concentration of parasite DNA as a measure of disease severity in falciparum malaria. J Infect Dis. 2015 Apr 1;211(7):1128-33. doi: 10.1093/infdis/jiu590. Epub 2014 Oct 24. PMID 25344520
- [Result] Pasricha SR, Atkinson SH, Armitage AE, Khandwala S, Veenemans J, Cox SE, Eddowes LA, Hayes T, Doherty CP, Demir AY, Tijhaar E, Verhoef H, Prentice AM, Drakesmith H. Expression of the iron hormone hepcidin distinguishes different types of anemia in African children. Sci Transl Med. 2014 May 7;6(235):235re3. doi: 10.1126/scitranslmed.3008249. PMID 24807559
- [Result] Hendriksen IC, White LJ, Veenemans J, Mtove G, Woodrow C, Amos B, Saiwaew S, Gesase S, Nadjm B, Silamut K, Joseph S, Chotivanich K, Day NP, von Seidlein L, Verhoef H, Reyburn H, White NJ, Dondorp AM. Defining falciparum-malaria-attributable severe febrile illness in moderate-to-high transmission settings on the basis of plasma PfHRP2 concentration. J Infect Dis. 2013 Jan 15;207(2):351-61. doi: 10.1093/infdis/jis675. Epub 2012 Nov 7. PMID 23136222
- [Result] Veenemans J, Schouten LR, Ottenhof MJ, Mank TG, Uges DR, Mbugi EV, Demir AY, Kraaijenhagen RJ, Savelkoul HF, Verhoef H. Effect of preventive supplementation with zinc and other micronutrients on non-malarial morbidity in Tanzanian pre-school children: a randomized trial. PLoS One. 2012;7(8):e41630. doi: 10.1371/journal.pone.0041630. Epub 2012 Aug 3. PMID 22870238
- [Result] Veenemans J, Milligan P, Prentice AM, Schouten LR, Inja N, van der Heijden AC, de Boer LC, Jansen EJ, Koopmans AE, Enthoven WT, Kraaijenhagen RJ, Demir AY, Uges DR, Mbugi EV, Savelkoul HF, Verhoef H. Effect of supplementation with zinc and other micronutrients on malaria in Tanzanian children: a randomised trial. PLoS Med. 2011 Nov;8(11):e1001125. doi: 10.1371/journal.pmed.1001125. Epub 2011 Nov 22. PMID 22131908
- [Result] Veenemans J, Jansen EJ, Baidjoe AY, Mbugi EV, Demir AY, Kraaijenhagen RJ, Savelkoul HF, Verhoef H. Effect of alpha(+)-thalassaemia on episodes of fever due to malaria and other causes: a community-based cohort study in Tanzania. Malar J. 2011 Sep 22;10:280. doi: 10.1186/1475-2875-10-280. PMID 21939508
- [Result] Veenemans J, Mank T, Ottenhof M, Baidjoe A, Mbugi EV, Demir AY, Wielders JP, Savelkoul HF, Verhoef H. Protection against diarrhea associated with Giardia intestinalis Is lost with multi-nutrient supplementation: a study in Tanzanian children. PLoS Negl Trop Dis. 2011 Jun;5(6):e1158. doi: 10.1371/journal.pntd.0001158. Epub 2011 Jun 7. PMID 21666789
- [Result] Mbugi EV, Meijerink M, Veenemans J, Jeurink PV, McCall M, Olomi RM, Shao JF, Chilongola JO, Verhoef H, Savelkoul HF. Effect of nutrient deficiencies on in vitro Th1 and Th2 cytokine response of peripheral blood mononuclear cells to Plasmodium falciparum infection. Malar J. 2010 Jun 14;9:162. doi: 10.1186/1475-2875-9-162. PMID 20546583
- [Result] Mbugi EV, Meijerink M, Veenemans J, Jeurink PV, McCall M, Olomi RM, Shao JF, Verhoef H, Savelkoul HF. Alterations in early cytokine-mediated immune responses to Plasmodium falciparum infection in Tanzanian children with mineral element deficiencies: a cross-sectional survey. Malar J. 2010 May 17;9:130. doi: 10.1186/1475-2875-9-130. PMID 20470442
- [Result] Veenemans J, Andang'o PE, Mbugi EV, Kraaijenhagen RJ, Mwaniki DL, Mockenhaupt FP, Roewer S, Olomi RM, Shao JF, van der Meer JW, Savelkoul HF, Verhoef H. Alpha+ -thalassemia protects against anemia associated with asymptomatic malaria: evidence from community-based surveys in Tanzania and Kenya. J Infect Dis. 2008 Aug 1;198(3):401-8. doi: 10.1086/589884. PMID 18582194